CLINICAL TRIAL: NCT02097381
Title: HIV Infection and Gut Mucosal Immune Function: Longitudinal Analyses of Intestinal CD4+ and Th17 T Cells in HIV-infected Individuals on Short-term Antiretroviral Therapy
Brief Title: Study of Recovery of Intestinal CD4+ and Th17 T Cells in HIV-infected Individuals on Short-term Antiretroviral Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Giancarlo Ceccarelli, MD, PhD, MSc, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DPHID-UniRoma01
Record Dates: First submitted 2014-03-17; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infection
Keywords: HIV infection; GUT; microbial translocation; chronic inflammation; antiretroviral therapy; cART; HAART; Th17; Th1; CD4+
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Darunavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- naïve for cART that met the criteria to start treatment (Other): patients naïve for antiretroviral treatment that met the criteria to start cART according to International Guidelines.
  These patients will be studied for primary and secondary outcomes after a short term antiretroviral therapy.
  Interventions: Drug: Tenofovir-Emtricitabine plus Lopinavir/Ritonavir or Darunavir/Ritonavir

INTERVENTIONS:
Drug: Tenofovir-Emtricitabine plus Lopinavir/Ritonavir or Darunavir/Ritonavir — Conventional antiretroviral therapy started in naïve patients for antiretroviral treatment that met the criteria to start cART according to International Guidelines.
  The antiretroviral treatment consisted in a tenofovir-emtricitabine NRTI backbone (TDF/FTC, 300/200 mg/ml, once a day) plus boosted protease inhibitor, lopinavir/ritonavir (LPV/r, 400/100 mg twice a day) or darunavir/ritonavir (DRV/r 800/100mg once a day).
  Other Names: Truvada; Prezista; Kaletra; Norvir

SUMMARY:
HIV infection is associated with a state of chronic, generalized immune activation that has been shown in many studies to be a key predictor of progression to AIDS. The molecular, cellular, and pathophysiological mechanisms underlying the HIV-associated immune activation are complex and still poorly studied. There is, however, growing consensus that both viral and host factors contribute to this phenotype, with emphasis on the role played by the mucosal immune dysfunction (and consequent microbial translocation). Moreover if it is known that in HIV-infected individuals, a severe depletion of intestinal cluster of differentiation 4 (CD4+) T-cells, is associated with loss of epithelium integrity, microbial translocation and systemic immune activation, the kinetics of intestinal CD4+ T-cell reconstitution under combined antiretroviral therapy (cART) remains poorly understood.

This study sought to evaluate the reconstitution of intestinal CD4+ T-cells, including Th1 and Th17, in blood and colon samples collected from HIV-infected individuals before and after a short term cART.

ELIGIBILITY:
Inclusion Criteria:

* naïve for antiretroviral treatment
* met the criteria to start cART according to International Guidelines
* written informed consent signed

Exclusion Criteria:

* treatment with glucocorticosteroids and any immune modulating medication for more than seven days in the previous month
* any past or current systemic malignancy, history of inflammatory diseases of the small or large intestine
* pregnancy
* anemia, use of anticoagulants, and any contraindications to phlebotomy or colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Difference of number of total Th1 and Th17 CD4+ T-cells (cell/mmc and %) in colon samples between T0 (before start of cARV) and T1 (after 6 months of cARV) | 6 months
  recovery of total Th1 and Th17 CD4+ T-cells (cell/mmc and %) in gut mucosa after 6 months of cARV)

SECONDARY OUTCOMES:
Difference of number of total Th1 and Th17 CD4+ T-cells (cell/mmc and %) in blood samples between T0 (before start of cARV) and T1 (after 6 months of cARV) | 6 months
  recovery of total Th1 and Th17 CD4+ T-cells (cell/mmc and %) in peripheral blood after 6 months of cARV)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Vullo, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Public Health and Infectious Diseases, University of Rome "Sapienza", Italy, Rome, RM, Italy

REFERENCES:
- [Derived] d'Ettorre G, Baroncelli S, Micci L, Ceccarelli G, Andreotti M, Sharma P, Fanello G, Fiocca F, Cavallari EN, Giustini N, Mallano A, Galluzzo CM, Vella S, Mastroianni CM, Silvestri G, Paiardini M, Vullo V. Reconstitution of intestinal CD4 and Th17 T cells in antiretroviral therapy suppressed HIV-infected subjects: implication for residual immune activation from the results of a clinical trial. PLoS One. 2014 Oct 23;9(10):e109791. doi: 10.1371/journal.pone.0109791. eCollection 2014. PMID 25340778